CLINICAL TRIAL: NCT05082766
Title: Improvement in the Appearance of Periorbital Wrinkles With DefenAge 8-in-1 BioSerum Supplemented With Enhanced Concentration of Defensins
Brief Title: Improvement in the Appearance of Periorbital Wrinkles
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: Advanced Dermatology (Other); MediCell Technologies, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DefenAge-2021-01
Record Dates: First submitted 2021-09-24; First posted 2021-10-19 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Periorbital Wrinkles
Keywords: wrinkles; crow's feet; face wrinkles; face; cosmetic
MeSH Terms: conditions — Facies

STUDY DESIGN:
Intervention Model Description: will be treated with the enhanced DefenAge 8-in-1 BioSerum to their entire face
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DefenAge 8-in-1 BioSerum supplemented with enhanced concentration of defensins (Experimental): Enrolled subjects will all receive enhanced DefenAge 8-in-1 BioSerum to be applied on the face including periorbital area.
  Interventions: Drug: enhanced DefenAge 8-in-1 BioSerum

INTERVENTIONS:
Drug: enhanced DefenAge 8-in-1 BioSerum — DefenAge is a topical skincare brand containing a composition of biologically active natural molecules, named defensins, that repair skin damage associated with aging.

SUMMARY:
The primary objective of this study is to evaluate the efficacy of DefenAge 8-in-1 BioSerum supplemented with the enhanced concentration of defensins (enhanced 8-in-1 BioSerum) in the improvement of periorbital wrinkles.

DETAILED DESCRIPTION:
Enrolled subjects will all receive enhanced DefenAge 8-in-1 BioSerum to be applied on the face including periorbital area.

Subjects satisfying all inclusion and exclusion criteria will be enrolled in this trial. Prior to receiving any study treatment, mandatory photography using Canfield Vectra 3D and VISIA. Patients will return for follow-up assessments at Day 30, 60, and 90.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects in general good health greater than 30 years of age
* Must be willing and capable of giving consent and signing an Informed Consent Form
* Subjects with moderate to severe periorbital wrinkles (at least a grade II in wrinkles and score of 4 in elastosis on the Fitzpatrick-Goldman wrinkle scale)
* Female Subjects will be either of non-childbearing potential defined as:

  1. Having no uterus
  2. No menses for at least 12 months
  3. Bilateral tubal ligation Or; (WOCBP) women of childbearing potential, must have had a regular menstrual cycle prior to study entry. All systemic birth control measures must be in consistent use at least 6 months prior to study participation. WOCBP must agree to use an effective method of birth control during the course of the study, such as:

  <!-- -->

  1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
  2. Intrauterine coil
  3. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
  4. Abstinence or same sex partner (If practicing abstinence or sexual activity with a same sex partner, must agree to use barrier method described above (c) if becomes sexually active with a non-vasectomized male partner).
  5. Vasectomized male partner (for at least 6 months) (must agree to use barrier method described above (c) if becomes sexually active with un-vasectomized male partner).
* Negative urine pregnancy test results at Baseline prior to study entry (if applicable)

Exclusion Criteria:

* History of sensitivity to any ingredient in DefenAge 8-in-1 BioSerum.
* Subjects receiving any topical cosmetic anti-wrinkle and/or skin lightening products known to affect skin aging such as products containing hydroquinone, vitamin A derivatives (retinol, tretinoin, adapalene, tazarotene), alpha/beta/poly-hydroxy acids (salicylic acid, glycolic acid etc.), vitamins C or D (includes derivatives thereof), arbutin, retinol, azelaic acid, kojic acid, licorice extracts, bearberry extracts, mequinol) on the treatment area within 14 days prior to or during the study period, other than the study product.
* Subjects using any topical imiquimod, 5-fluorouracil, or diclofenac on their face within 12 weeks prior to or during the study period
* Subjects who have had a microdermabrasion (light or medium skin peel on their face within 30 days prior to or during the study period
* Subjects receiving a chemical peel, a non-ablative laser, light, radiofrequency, or ultrasound treatment on their face must have discontinued the drug/treatment at least 3 months prior to entering the study
* Subjects receiving Dermabrasion (deep skin peel) and/or ablative laser treatments on their face, and systemic retinoids must have discontinued the drug/treatment at least 6 months prior to entering the study
* History of or the presence of any skin condition/disease that might, in the opinion of the investigator, interfere with the diagnosis or evaluation of study parameters (i.e., acne, atopic dermatitis, eczema, psoriasis, seborrheic dermatitis)
* Subjects with current actinic keratoses or any other skin cancer(s) in the treatment areas
* Subjects with a significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would preclude enrollment into the study
* Subjects with any active systemic disease that is not yet deemed medically stabilized
* Subjects with an active bacterial, fungal, or viral infection
* Subjects participating or completing participation in a clinical trial within 30 days prior to or during the study period
* A female subject who is currently breast-feeding, nursing, pregnant or planning to becoming pregnant during the study period
* Subjects not willing to comply with study dosing and complete the entire course of the study
* Subjects not willing to avoid extended periods of sun exposure for the duration of the study (including tanning beds). During the study, when excessive sun exposure is unavoidable, subjects should wear appropriate protective clothing and use the dispersed sunscreen
* Subjects who have had treatment with neuromodulators (ex. Botox, Dysport, or Xeomin) anywhere on the face within 6 months prior to or during the study period.

  18. Subjects who have had treatment with fillers anywhere on the face, or other forms of facial soft tissue augmentation (ex. Fat transfer) within 6 months prior to or during the study period.

Min Age: 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-10-11 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinician evaluator assessment of change using Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale | baseline, Day 30, Day 60, and Day 90
  measurements will be completed based on images captured at baseline, Day 30, Day 60, and Day 90 and assessed by a blinded evaluator using the Fitzpatrick-Goldman Classification of Wrinkling and Degree of Elastosis Scale where wrinkling ranges from class 1 (fine wrinkles) to class 3 (Fine to deep wrinkles, numerous lines, with or without redundant skin folds) and Elastosis ranges from 1-3 (mild) to 7-9 (severe)
Asses the change of Percent of improvement at different time points | Day 30, Day 60, and Day 90
  Percent improvement in periorbital wrinkles, laxity, pigmentation, erythema, texture, and radiance conducted by an evaluator

SECONDARY OUTCOMES:
Investigator-assessed Global Aesthetic Improvement Score (I-GAIS) | Day 30, 60 and 90
  Investigator-assessed Global Aesthetic Improvement Score based on photographs where scale is 1 (much improved) to 5 (much worse)
Subject Global Aesthetic Improvement Score (S-GAIS) | Day 30, 60 and 90
  Subject Global Aesthetic Improvement Score Day 30, 60 and 90 using photographs where scale is 1 (much improved) to 5 (much worse)
Investigator assessment of tolerability of study drug including erythema, burning/stinging, dryness, peeling (desquamation), and tenderness | Day 30, 60 and 90.
  Investigator assessment of tolerability of study drug
Patient questionnaire | Day 30, 60 and 90.
  Self-Assessment questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina G Fabi, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- West Dermatology Research Center/Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Possibly Efficacy Data-endpoints

REFERENCES:
- [Background] Taub A, Bucay V, Keller G, Williams J, Mehregan D. Multi-Center, Double-Blind, Vehicle-Controlled Clinical Trial of an Alpha and Beta Defensin-Containing Anti-Aging Skin Care Regimen With Clinical, Histopathologic, Immunohistochemical, Photographic, and Ultrasound Evaluation. J Drugs Dermatol. 2018 Apr 1;17(4):426-441. PMID 29601620